CLINICAL TRIAL: NCT05913778
Title: Long-term Effects of Enhanced External Counterpulsation on the Structural and Functional State of Blood Vessels in Patients With Coronary Heart Disease and Chronic Heart Failure
Brief Title: Long-tErm Effects of Enhanced eXternal CountErpuLsation
Acronym: EXCEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUCT10122020
Record Dates: First submitted 2023-06-01; First posted 2023-06-22 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-10

CONDITIONS: Coronary Artery Disease; Chronic Heart Failure
Keywords: coronary artery disease; chronic heart failure; enhanced external counterpulsation; structural and functional vascular state; clinical status; exercise tolerance; quality of life; cardiovascular events
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: open, prospective, randomized, controlled in parallel groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Enhanced external counterpulsation 35 hours per year (Experimental): Subjects with Heart failure with Enhanced external counterpulsation therapy (inflation pressure 220-280 mm Hg; 35 procedures) was given as a 1-hour session, once daily, for a total of 35 sessions, 1 course per 12 months
  Interventions: Device: Enhanced external counterpulsation
- Enhanced external counterpulsation 70 hours per year (Experimental): Subjects with Heart failure with Enhanced external counterpulsation therapy (inflation pressure 220-280 mm Hg; 35 procedures) was given as a 1-hour session, once daily, for a total of 35 sessions, 1 course per 6 months
  Interventions: Device: Enhanced external counterpulsation
- SHAM external counterpulsation (Sham Comparator): Subjects with Heart failure with SHAM external counterpulsation (inflation pressure 80 mm Hg; 35 procedures) was given as a 1-hour session, once daily, for a total of 35 sessions, 1 course per 12 months
  Interventions: Device: Enhanced external counterpulsation

INTERVENTIONS:
Device: Enhanced external counterpulsation — Enhanced external counterpulsation (EECP) is a noninvasive therapy for the treatment of patients with coronary artery disease.The systolic deflation/diastolic inflation sequence of EECP leads to systolic unloading and diastolic augmentation, resulting in increased blood flow in a pulsatile manner in coronary artery and in others organ arteries.
  Other Names: EECP

SUMMARY:
Enhanced external counterpulsation (EECP) is an effective non-invasive treatment in patients with coronary artery disease (CAD) which complicated by chronic heart failure (CHF).

Aim: to study the long-term effects of treatment with enhanced external counterpulsation on the structural and functional state of the vascular bed in patients with stable CAD complicated by CHF.

Patients (n=100) with verified stable CAD (class 2-3 angina) complicated by CHF (NYHA class 2-3) and receiving optimal drug therapy included in open randomized study.

Primary randomization (2:1) + secondary randomization (1:1).

* SHAM-counterpulsation group (ECP-SHAM; compression pressure 80 mm Hg; 35 procedures, 1 hour each);
* Active counterpulsation group (ECP35; compression pressure 220-280 mm Hg; 35 procedures, 1 hour each) 1 course per year;
* Active counterpulsation group (ECP70; compression pressure 220-280 mm Hg; 35 procedures, 1 hour each) 2 courses per year.

Duration of observation is 3 years. Stages of examination: after 3, 6, 12, 24, 36 months (after 3, 6, 12 months for the ECP-SHAM group).

Primary endpoint: combination of vascular event (myocardial infarction, acute cerebrovascular accident, revascularization procedures), hospitalization (for CAD/CHF), death.

Secondary endpoints: changes in exercise tolerance, a needing for antianginal therapy, frequency of angina episodes.

Objectives: to study the dynamics of the structural and functional state of the vascular bed (applanation tonometry, photoplethysmography, computer nailfold videocapillaroscopy), the dynamics of the clinical status (Clinical Status Assessment Scale), the dynamics of exercise tolerance (6-minute walk test), the dynamics of the quality of life of patients ( questionnaires SF36 and MLHFQ) in the ECP35 and ECP70 groups at baseline, at the end of the first course, after 6 months, 1, 2, and 3 years, and in the ECPSHAM group at baseline, at the end of the first course, after 6 and 12 months; (2) To investigate the impact of EECP on the incidence of primary (vascular events, hospitalizations for CAD/CHF, death) and secondary (frequency of angina episodes, need for antianginal drugs, exercise tolerance) endpoints.

Expected outcome of the study: Obtaining reliable data on the long-term positive effect of EECP on the dynamics of the structural and functional state of the vascular bed, exercise tolerance, quality of life and prognosis in patients with stable CAD complicated by CHF.

DETAILED DESCRIPTION:
1. Topic relevance

   The dominant positions of coronary artery disease (CAD) in the structure of morbidity, disability and mortality among patients with cardiovascular diseases determine the social significance of this disease. With an increase in the incidence of cardiovascular diseases from 2.483 million cases in 2000 to 4.784 million cases in 2018 (an increase of 193%), there is also an increase in newly diagnosed cases of CAD by 47%. The mortality rate from circulatory diseases in Russia over the past 15 years has decreased from 927.5 to 587.6 per 100,000 population. Achievements of modern medicine (optimization of pharmacotherapy and an increase in the number of revascularization procedures) have contributed to an improvement in the survival rates of patients with CAD. However, with an increase in life expectancy, the economic burden of atherosclerotic diseases and the need to improve the quality of life of such patients increase.

   Taking into account the insufficient effect of a conservative strategy in patients with severe stenoses in the coronary bed, a clear increase in the number of revascularization procedures has been observed over the past two decades. However, the limited duration of the effective functioning of stents and shunts, as well as the lack of proven benefits in terms of influencing the prognosis compared to conservative measures do not allow to fully rely on this strategy as well. In the population, there is an accumulation of the proportion of people with refractory angina pectoris, with insufficient effectiveness of the use of conservative and invasive strategies. The basis of this population is patients with progression of multivessel coronary atherosclerosis, microvascular disease, incomplete myocardial revascularization, stenosis or occlusion of shunts / stents, and patients who cannot undergo coronary bypass surgery or stenting, including repeated ones, for various other reasons. In addition, the course of coronary artery disease in such patients is often complicated by chronic heart failure (CHF), which further reduces the quality of life of patients and the prognosis. This determines the search for additional methods of treatment for these patients, which can enhance the effect of conservative and invasive strategies.

   Enhanced external counterpulsation (EECP) is an effective non-invasive and atraumatic treatment for patients with coronary artery disease, including complicated CHF. Preference should be given to this method in patients with severe diffuse lesions of the coronary arteries, in case of impossibility or high risk of myocardial revascularization, as well as in case of complication of heart failure. The influence of this method on the contractility of the heart, exercise tolerance and quality of life of these patients has been studied quite well. However, the long-term effects of EECP on the structural and functional state of the vascular bed (the main targets of this method) in patients with coronary artery disease complicated by CHF remain little studied.
2. The novelty of the proposed topic on literary sources and patent documentation. No similarly designed studies were found in the available literature. Scientific novelty It is planned to study long-term vascular effects, the impact on exercise tolerance, quality of life, the frequency of serious adverse events, the impact on the prognosis during the treatment of EECP patients with stable CAD complicated by CHF. It is planned to expand the possible indications for EECP, optimize the treatment of EECP in patients with refractory angina and heart failure.
3. Purpose and objectives of the planned research. Purpose of the study - To study the long-term effects of treatment with EECP on the structural and functional vascular state in patients with stable CAD complicated by CHF.

   Research objectives.

   • To study the dynamics of the structural and functional vascular state (applanation tonometry, photoplethysmography, computer nailfold capillaroscopy) in active EECP groups (220-280 mm Hg; 35 procedures) 2 courses per year or 1 course per year initially, according to at the end of the course, after 6 months, 1, 2 and 3 years and in the SHAM external counterpulsation group (placebo; 80 mm Hg; 35 procedures) at baseline, at the end of the course, after 6 and 12 months;

   • To study the dynamics of the clinical status (Clinical State Assessment Scale) in the groups of active EECP (220-280 mm Hg; 35 procedures) 2 courses per year or 1 course per year initially, at the end of the course, after 6 months, 1, 2 and 3 years and in the SHAM external counterpulsation group (placebo; 80 mm Hg; 35 procedures) at baseline, at the end of the course, after 6 and 12 months;

   • To study the dynamics of exercise tolerance (6-minute walk test) in active EECP groups (220-280 mm Hg; 35 procedures) 2 courses per year or 1 course per year initially, at the end of the course, after 6 months, 1, 2 and 3 years and in the SHAM external counterpulsation group (placebo; 80 mm Hg; 35 procedures) at baseline, at the end of the course, after 6 and 12 months;
   * To study the dynamics of the quality of life of patients (SF36 and MLHFQ questionnaires) in the groups of active EECP (220-280 mm Hg; 35 procedures) 2 courses per year or 1 course per year through the baseline, at the end of the course, 6 months, 1 , 2 and 3 years and in the SHAM external counterpulsation group (placebo; 80 mm Hg; 35 procedures) at baseline, at the end of the course, after 6 and 12 months;
   * To study the dynamics of the frequency of angina pectoris episodes, the need for antianginal drugs, the frequency of vascular events, hospitalizations (for coronary artery disease / CHF), deaths in active EECP groups (220-280 mm Hg, 35 procedures) for 2 or 1 course per year and in the SHAM external counterpulsation group (placebo; 80 mm Hg; 35 procedures) during the observation period.
   * To study the effect of EECP on the incidence of primary (vascular events, hospitalizations for CAD/CHF, deaths) and secondary (frequency of angina episodes, need for antianginal drugs, exercise tolerance) endpoints;
   * Perform a correlation analysis between EECP treatment parameters (number of procedures and duration of treatment) with the characteristics under study (vascular and clinical effects).
4. Planned type of scientific research The study is open, prospective, randomized, controlled in parallel groups.
5. Object of study and the planned number of observations. The object of the study were patients (n=100) with verified CAD (class 2-3, stable angina), complicated by CHF (NYHA class 2-3), receiving optimal drug therapy.

Inclusion Criteria:

* Age 40-75 years
* Verified CAD (class 2-3, stable angina) complicated by CHF (NYHA class 2-3)
* Signed voluntary informed consent to participate in the study

Non-inclusion/exclusion criteria:

* Contraindications to treatment with EECP: recent (2-4 weeks ago) catheterization of arterial vessels; cardiac arrhythmias that can affect the synchronization of counterpulsation with the ECG; decompensated heart failure; left ventricular ejection fraction less than 30%; severe aortic insufficiency; critical ischemia of the arteries of the lower extremities; thrombosis / thrombophlebitis of the veins of the lower extremities; uncontrolled arterial hypertension (>180/110mm Hg); high pulmonary hypertension (grade 2-3; >45 mm Hg); coagulopathy, treatment with anticoagulants with prothrombin time >15 sec/INR >3; pregnancy; aneurysm of the thoracic or abdominal aorta requiring surgical treatment.
* Refusal of the patient from further participation in the study.

  6. Specific methods of the planned research

  (1) Clinical analysis of present symptoms. (2) General clinical examination, including laboratory research methods (general blood count, general urinalysis, biochemical blood test) and instrumental studies (electrocardiography, echocardiography, daily ECG monitoring, ultrasound of the vessels of the lower extremities).

  (3) Assessment of exercise tolerance (6-minute walk test). (4) Evaluation of the functional status (Scale for Assessment of the Clinical State as modified by V.Yu. Mareev).

  (5) Quality of life assessment: Questionnaire SF-36 (The Short Form-36); MLHFQ (Minnesota Living With Heart Failure Questionnaire; Minnesota Living With Heart Failure Questionnaire).

  (6) Non-invasive vascular examination: assessment of remodeling of the microvasculature: computer nailfold capillaroscopy (Capillaroscan-1, Russia); determination of the structural and functional state of the walls of large vessels and microvasculature: photoplethysmography (Angioscan-01, Russia); determination of the level of central arterial pressure, augmentation index: applanation tonometry (A-pulse CASPro, USA).

  (7) The study of patients' self-monitoring diaries (frequency of angina episodes, need for antianginal drugs), the frequency of hospitalizations for coronary artery disease/CHF, the frequency of vascular events/revascularizations.

  7. The expected result of the study. Obtaining reliable data on the long-term positive effect of EECP on the dynamics of the structural and functional vascular state, exercise tolerance, quality of life and prognosis in patients with stable CAD complicated by CHF. To substantiate the wider inclusion of treatment with EECP in a comprehensive program for the management of patients with CAD, including complicated CHF, along with a conservative and invasive strategy, to optimize the treatment with EECP in these patients. Presentation of the results obtained in the form of publications and implementation of the results in practical healthcare (expansion of indications for the treatment of EECP; reference to training programs for doctors).

  8. Base of scientific research. Department of Hospital Therapy No. 1, First Moscow State Medical University. THEM. Sechenov (University Clinical Hospital No. 1, First Moscow State Medical University named after I.M. Sechenov).

  9. Calendar terms of performance of work:
  1. Beginning of material collection December 2020
  2. Completion of the collection of material December 2021

ELIGIBILITY:
Inclusion Criteria:

* Age 40-75 years
* Verified CAD (class 2-3, stable angina) complicated by CHF (NYHA class 2-3)
* Optimal medical treatment
* Signed voluntary informed consent to participate in the study

Exclusion Criteria:

* Contraindications to treatment with EECP: recent (2-4 weeks ago) catheterization of arterial vessels; cardiac arrhythmias that can affect the synchronization of counterpulsation with the ECG; decompensated heart failure; left ventricular ejection fraction less than 30%; severe aortic insufficiency; critical ischemia of the arteries of the lower extremities; thrombosis / thrombophlebitis of the veins of the lower extremities; uncontrolled arterial hypertension (>180/110mm Hg); high pulmonary hypertension (grade 2-3; >45 mm Hg); coagulopathy, treatment with anticoagulants with prothrombin time >15 sec/INR >3; pregnancy; aneurysm of the thoracic or abdominal aorta requiring surgical treatment.
* Refusal of the patient from further participation in the study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Composite primary endpoint | 12 months, 24 months, 36 months
  combination of vascular event (myocardial infarction, acute cerebrovascular accident, revascularization procedures), hospitalization (for CAD/CHF), death

SECONDARY OUTCOMES:
Exercise tolerance | 3 months, 6 months, 12 months, 24 months, 36 months
  changes in exercise tolerance (6-minute walk test)
Antianginal therapy | 12 months, 24 months, 36 months
  changes in need for antianginal therapy (nitroglycerin doses per week)
Angina episodes | 12 months, 24 months, 36 months
  changes in frequency of angina episodes

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Lishuta, MD, PhD, Principal Investigator — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (1):
- I.M. Sechenov First Moscow State Medical University (Sechenov University), Moscow, Russia

REFERENCES:
- [Background] Karaganov K.S., Lishuta A.S., Belenkov Y.N. The Use of Enhanced External Counterpulsation in the Treatment of Patients with Coronary Artery Disease. Rational Pharmacotherapy in Cardiology. 2020;16(4):579-584. (In Russ.) https://doi.org/10.20996/1819-6446-2020-08-07
- [Background] Karaganov K.S., Slepova O.A., Lishuta A.S., Solomakhina N.I., Belenkov Yu.N. Medium-term Effects of Enhanced External Counterpulsation in the Structural and Functional Parameters of Blood Vessels in Patients with Coronary Artery Disease. Rational Pharmacotherapy in Cardiology. 2021;17(4):557-563. https://doi.org/10.20996/1819-6446-2021-08-03
- [Background] Slepova O.A., Lishuta A.S., Vasiltsova E.Yu., Privalova E.V., Belenkov Yu.N. The Effect of Enhanced External Counterpulsation on the Vascular State, Indicators of Glycemic Control and Quality of Life in Patients with Coronary Artery Disease and Type 2 Diabetes Mellitus. Rational Pharmacotherapy in Cardiology. 2022;18(3):274-281. https://doi.org/10.20996/1819-6446-2022-06-04
- [Background] Mamieva Z.A., Lishuta A.S., Belenkov Yu.N., Privalova E.V., Yusupova A.O., Rykova S.M. POSSIBILITIES OF ENHANCED EXTERNAL COUNTERPULSATION USING IN CLINICAL PRACTICE. Rational Pharmacotherapy in Cardiology. 2017;13(2):238-247. (In Russ.) https://doi.org/10.20996/1819-6446-2017-13-2-238-247
- [Result] Lishuta A.S., Nikolaeva N.A., Belenkov Yu.N. Long-term vascular effects of enhanced external counterpulsation in patients with coronary artery disease complicated by heart failure. Medical and pharmaceutical journal "Pulse". 2024; 26 (4): 81-89. http://dx.doi.org//10.26787/nydha-2686-6838-2024-26-4-81-89
- [Result] Lishuta A.S., Slepova O.A., Nikolaeva N.A., Belenkov Yu.N. Medium-term effects of enhanced external counterpulsation on markers of glycemic control in patients with chronic heart failure of ischemic genesis. Medical and pharmaceutical journal "Pulse". 2024; 26 (5): 92-99. http://dx.doi.org//10.26787/nydha-2686-6838-2024-26-5-92-99
- [Result] Lishuta A.S., Nikolaeva N.A., Belenkov Yu.N. Long-term effectiveness of enhanced external counterpulsation in patients with chronic heart failure of ischemic genesis. Medical and pharmaceutical journal "Pulse". 2024; 26 (6): 63-70. http://dx.doi.org//10.26787/nydha-2686-6838-2024-26-6-63-70
- [Result] Lishuta A.S., Slepova O.A., Nikolaeva N.A., Privalova E.V., Belenkov Yu.N. Long-term effects of enhanced external counterpulsation in the management of patients with coronary artery disease complicated by heart failure: data from the EXCEL study. Creative cardiology. 2024; 18 (2): 194-201. DOI: 10.24022/1997-3187-2024-18-2-194-201
- [Result] Belenkov YN, Lishuta AS, Slepova OA, Nikolaeva NS, Khabarova NV, Dadashova GM, Privalova EV. The EXCEL Study: Long-term Observation of the Effectiveness of Drug and Non-drug Rehabilitation in Patients with Ischemic Heart Failure. Kardiologiia. 2024 Jan 31;64(1):14-24. doi: 10.18087/cardio.2024.1.n2615. English, Russian. PMID 38323440
- [Result] Lishuta A.S., Slepova O.A., Nikolaeva N.A., Khabarova N.V., Privalova E.V., Belenkov Yu.N. Effectiveness of different treatment regimens of enhanced external counterpulsation in patients with stable coronary artery disease complicated by heart failure. Rational Pharmacotherapy in Cardiology. 2024;20(1):35-45. https://doi.org/10.20996/1819-6446-2024-3004.
- [Result] Lishuta A.S., Slepova O.A., Nikolaeva N.A., Petruhnova M.F., Privalova E.V., Belenkov Yu.N. Long-term effects of enhanced external counterpulsation in the management of patients with ischemic chronic heart failure. Rational Pharmacotherapy in Cardiology. 2024;20(2):194-201. https://doi.org/10.20996/1819-6446-2024-3041
- [Result] Lishuta A.S., Slepova O.A., Nikolaeva N.S., Privalova E.V., Belenkov Yu.N. Long-term effects of enhanced external counterpulsation in the management of patients with coronary artery disease complicated by heart failure: data from the EXCEL study. Russian Journal of Cardiology. 2024;29(6):5886. https://doi.org/10.15829/1560-4071-20245886.
- [Result] Lishuta A.S., Privalova E.V., Belenkov Yu.N. Enhanced external counterpulsation in the management of patients with ischemic heart failure: long-term impact on clinical outcomes. Cardiovascular Therapy and Prevention. 024;23(8):4015. https://doi.org/10.15829/1728-88002024-4015